CLINICAL TRIAL: NCT02721394
Title: Conducting Functional Communication Training (FCT) With Young Children With Intellectual Disabilities in NHS Settings in the UK: A Feasibility Project
Brief Title: FCT With Young Children With ID in the UK: A Feasibility Project V.1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Kent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ResGov 325
Record Dates: First submitted 2016-02-29; First posted 2016-03-29 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Intellectual Disability
Keywords: Challenging Behaviour; Functional Communication Training; Positive Behavioural Support; Family carer training
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Researcher Implemented FCT (Experimental): Children receive functional communication training. Assessment and initial intervention sessions are completed by the researcher and family carers are trained to continue the intervention at home.
  Interventions: Behavioral: Functional Communication Training
- Family Carer Implemented FCT 1 (Experimental): Children receive functional communication training. Family carers are trained to implement all sessions (including assessment and initial intervention sessions) with coaching from the researcher in person.
  Interventions: Behavioral: Functional Communication Training
- Family Carer Implemented FCT 2 (Experimental): Children receive functional communication training. Family carers are trained to implement all sessions (including assessment and initial intervention sessions) with coaching from the researcher via videoconferencing and support from a family carer assistant in person.
  Interventions: Behavioral: Functional Communication Training

INTERVENTIONS:
Behavioral: Functional Communication Training — Functional Communication Training (which aims to teach the child a communicative alternative to challenging behaviour) implemented by either the researcher or family carer.

SUMMARY:
The current project aims to assess the feasibility of conducting Functional Communication Training in the UK with a small sample of young children (aged under 9) in an NHS setting. Three delivery formats will be assessed in order to demonstrate the feasibility of conducting FCT via different delivery methods within an NHS context. Participants will be four children aged under 9 who have an identified intellectual / developmental disability and display either self-injury, property destruction, or aggression at home. In addition, one family carer per child will be coached to implement the intervention, either following researcher intervention, or from the beginning. Data will be collected on challenging behaviour, communication responses, family carer confidence in managing behaviour, fidelity of intervention implementation, family quality of life, and acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child aged under 9
* Child has identified intellectual disability or genetic syndrome associated with intellectual disability (e.g. Fragile X Syndrome)
* Child uses only phrase speech (i.e. 2-3 word utterances)
* Child displays self injury, aggression, property destruction at home
* Family carers aged over 18 with capacity to consent
* Family carer speaks English as first language (to ensure that the child understands English and will therefore understand researcher)

Exclusion Criteria:

* Child experiences health condition involving pain that is not well controlled by treatment
* Child is fully deaf / blind
* Child or family carer receiving active treatment in relation to child's behaviour (e.g. direct behavioural support, parenting programme etc.)

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Observation of frequency or duration challenging behaviour | During functional analysis (2 sessions), intervention (4 sessions), maintenance (3 sessions) & follow up (1 session). Across a total of approximately 6 months.
  Observational measure of the frequency or duration of child target behaviours. This measure is expected to show a change over time as the intervention progresses, therefore data is collected during every session.

SECONDARY OUTCOMES:
Observation of occurrence of communication | During intervention (4 sessions), maintenance (3 sessions), & follow up (1 session). Across a total of approximately 5 months.
  Observational measure of the frequency of the child's use of the alternative communication response. This measure is expected to show a change over the course of the intervention and data will therefore be collected during each session.
Beech Centre Family Quality of Life Scale (Park et al., 2003) | At beginning of study, immediately after intervention (approximately 6-8 weeks later), and at final follow up session (approximately 6 months after beginning of the study).
  Questionnaire evaluating family quality of life. This measure is expected to show a change over time as the intervention progresses, therefore data is collected at 3 time points (pre intervention, post intervention, and at final follow up).
Rating scale measuring intervention fidelity | During intervention sessions (4 sessions), maintenance sessions (3 sessions), and during follow up (1 session). Across a total of approximately 5 months.
  Individualised rating scales assessing fidelity of researcher or family carer implementation of the intervention.
Modified Challenging Behaviour Checklist (Harris, Humphreys, & Thomson, 1994) | At beginning of study, immediately after intervention (approximately 6-8 weeks later), and at final follow up session (approximately 6 months after beginning of the study).
  Questionnaire to assess changes in non-targeted behaviours. This measure is expected to show a change over time as the intervention progresses, therefore data is collected at 3 time points (pre intervention, post intervention, and at final follow up).
Functional Assessment Interview Communication Section (O'Neill, Albin, Storey, Horner, & Sprague, 2014) | At beginning of study, immediately after intervention (approximately 6-8 weeks later), and at final follow up session (approximately 6 months after beginning of the study).
  Questionnaire used to assess changes in non-targeted areas of communication. This measure is expected to show a change over time as the intervention progresses, therefore data is collected at 3 time points (pre intervention, post intervention, and at final follow up).
Modified Parenting Task Checklist (Sanders & Woolley, 2001; 2005) | At beginning of study, immediately after intervention (approximately 6-8 weeks later), and at final follow up session (approximately 6 months after beginning of the study).
  Questionnaire to assess family carer confidence in doing a range of activities with their child. This measure is expected to show a change over time as the intervention progresses, therefore data is collected at 3 time points (pre intervention, post intervention, and at final follow up).

OTHER OUTCOMES:
Treatment Acceptability Rating Form - Revised (Reimers & Wacker, 1988) | At final follow up session approximately 6 months after the beginning of the study.
  Questionnaire assessing the acceptability of the intervention to family carers.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - East Kent Hospitals University NHS Foundation Trust, Canterbury, Kent
  - Mencap Northern Ireland, Belfast

IPD SHARING:
Plan to Share IPD: No